CLINICAL TRIAL: NCT03381378
Title: Analysis of Associations Between s-25OHD and Hand Grip Strength at 5 Years in Odense Child Cohort
Brief Title: Vitamin D and Hand Grip Strength at 5 Years in Odense Child Cohort
Acronym: VITHGS
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Christesen, Consultant, Professor, MD, PhD, Odense University Hospital
Other Study IDs: VITHGS
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Hypovitaminosis D; Hand Grasp; Children
Keywords: Vitamin D; s-25-hydroxyvitamin D; hand grip strength; myopathy; muscle
MeSH Terms: conditions — Vitamin D Deficiency; Muscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Venous blood samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will encompass an analysis of an eventual association between vitamin D status (maternal during pregnancy, at birth or at 5 years) and hand grip strength at 5 years in children from Odense Child Cohort. Odense Child Cohort is a large-scale, prospective, population-based, follow-up study. Mothers and their children born from January 2010 to December 2012 and resident in the Municipality of Odense, Denmark, are followed from early pregnancy up to adulthood. Data is obtained from questionnaires and medical records and venous blood samples were drawn and stored at a biological bank.

Low muscle strength in children has been linked to adiposity, cardiovascular disease and metabolic risk factors and low muscle strength in adolescence has been shown to be a risk factor of early adulthood mortality. There are not many studies on muscle strength in small children. There is some evidence of vitamin D concentrations in the blood having a positive correlation to upper body muscle strength in adolescent girls.

Hypovitaminosis D defined as serum 25-hydroxyvitamin D <50nmol/L was evident in 27,8% of the pregnant women and 47,7% of the new-born children in Odense Child Cohort.

Animal studies have shown an effect of vitamin D on regulation of muscle function and development. Studies on humans adults have shown that vitamin D deficiency can lead to myopathy. Myopathy in children as a result of hypovitaminosis D is not well-studied.

Given the high prevalence of hypovitaminosis D, mild or severe vitamin D-associated myopathy may be prevalent in preschool children.

The objectives of this study are 1) to create reference values and determine predictors of hand grip strength at five years, 2) to analyze the associations between vitamin D at different time points and hand grip strength at 5 years.

DETAILED DESCRIPTION:
Background The hand grip test has previously been used to study muscle strength in children (1). The test has also been found to be a reliable alternative in population-based studies to the gold standard isokinetic dynamometry (2).

There is not much research on hand grip strength in preschoolers and no consensus about which variables explain the variance in the normal distribution (3-5).

S-25-hydroxyvitamin D (s-25OHD) <50 nmol/L is prevalent in Denmark particularly in the winter due to the lack of ultraviolet B exposure and insufficient dietary intake (6). Vitamin D deficiency can lead to vitamin D-associated myopathy before developing actual bone disease (7). Little is known about vitamin-D-associated myopathy in children. Given the high prevalence of hypovitaminosis D, vitamin D-associated myopathy may be prevalent in preschool children.

The main objectives of this study were to: 1) establish a normative data-set of hand grip measurements for five-year-old children and determine which variables (during pregnancy, at birth and current) are associated to hand grip strength at five years of age and 2) investigate the association between vitamin-D-status (at 5 years, at birth, in early and in late pregnancy) and hand grip strength at the age of five.

Methods As many 5-year old children from Odense Child Cohort (OCC)as possible will be included during the study period (January 2016-June 2017). Expected number of children investigated by study completion is 1200. The exclusion criteria are multiple birth, preterm birth (GA<259 days), chronic disease and missing hand grip data at five years.

Questionnaires, blood samples for s-25OHD analysis and examinations of height, weight, skinfold thickness and 5-year hand grip measurement data will be needed for this study. When available, questionnaire data will be validated using medical records.

Blood samples Blood samples were obtained from mothers during early and late pregnancy, from offspring cord at birth and from the children at 5-years. The blood samples were stored at -80o C. S-25(OH)D2+3 analyses will be performed by liquid chromatography mass spectrometry (LC-MS/MS) as previously described (8, 9)

Explanatory Variables Child sex, age, height, weight, Body mass index (BMI), triceps skinfold and subscapular skinfold will be examined as continuous variables and examination season, vitamin D supplements, parents' education, ethnicity, mother's parity, smoking during pregnancy, birth weight, birth length, organized sports, physical activity compared to peers, motor skills compared to peers and child choice of free time activities as categorical variables.

Primary association The primary exposure is 5-year s-25OHD and the primary outcome is hand grip strength at five years. A Sub-analysis split by sex will be done.

Other associations

* S-25OHD in early and late pregnancy and chord s-25OHD and hand grip.
* Prediction of myopathy defined as hand grip <10th percentile vs. >10th percentile.

Statistics:

Descriptive statistics for baseline data, exposures and outcomes will be presented as mean (standard deviation) for parametric data and median (inter-quartile range) for non-parametric data. The students t-test for parametric and Mann-Whitney test for non-parametric data will be used to test the differences between the sexes and the difference between participants and non-participants. Univariate and multivariate regression models will be used to analyze the obtained data and to control for co-variates affecting the associations. Multiple regression variables will be decided upon based on appearance in the existing literature and a univariate p-value <0.10 will determine addition of further variables. All data will be investigated in total and for each of the sexes separately. Linear models will be used to predict hand grip strength and logistic regression will be used to assess myopathy defined as hand grip <10th percentile vs. >10th percentile. S-25OHD will be investigated both as a continuous and as a categorical parameter split by quartiles and the routine cut offs 25, 50 and 75 nmol/L. Model goodness-off-fit will be checked for all final models. Likelihood ratio test will be used to assess interaction between sex and all other variables and between s-25OHD and other variables in the models. In case of missing data, models will be reanalyzed with complete data of variables in larger models. A p-value <0.05 will be considered significant and p<0.10 will be considered a trend. Power calculation (primary outcome): Expected N=1200, 1 SD hand grip 18.4 N, 1SD of s-25OHD 22 nmol/L, alpha=0.05 and beta=0.80. It is calculated that our study will be able to detect a true difference of 0.68 N per 10 nmol/L change in s-25OHD (univariate association).

Ethics The OCC vitamin D project is an observational study, carried out according to the Helsinki II declaration and approved by the Regional Scientific Ethical Committee for Southern Denmark, no. S-20090130 and the Danish Data Protection Agency, no. 16/42833. Hand grip examination is an already approved part of the standard examination of 5-y children in OCC as part of the vitamin D project. All parents signed consent forms to receive information and invitations to follow-up examinations from OCC. Both parents' and children's permissions will be obtained before blood is drawn at five years and the children will be free to refuse any part of the examinations.

ELIGIBILITY:
Inclusion Criteria:

* 5-year-old children participating in Odense Child Cohort.

Exclusion Criteria:

* Multiple and/or preterm birth (gestational age (GA) <259 days)
* Chronic disease
* No available hand grip data at five years.

Ages: 5 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study was conducted using data from the Odense Child Cohort. Mothers and their children born from January 2010 to December 2012 and resident in the Municipality of Odense, Denmark, were followed from early pregnancy up to five years at present. Approximately 2500 children were included.
Sampling Method: Non-Probability Sample
Enrollment: 881 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Hand Grip Strength at 5 years | Examination within a week of 5 year birthday. 3-5 measurements with a duration of 5 seconds each of each hand.
  DHD-1 Digital Hand Dynamometer is used to measure 5-year-old children's hand grip strength. According to standard protocol the child is instructed to hold the dynamometer and the handle is adjusted to the child's hand. The child must be able to press the handle using the whole hand and not just the finger joints. The child must sit with a straight back and feet on the ground. The arm must not be supported by the hip, the elbow must be flexed to 90 degrees and the hand must be in the natural position.
  The child is instructed to press as hard as possible but in a slow movement to avoid sudden changes in position that might affect the results. Each measurement is approximately 5 seconds long with 1 minute break in between measuring the right and left hand interchangeably. Three measurements of each hand are taken starting with the right hand. If the last measure is the highest, a fourth measurement is taken and a fifth and last measurement is taken if the fourth is the highest.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stark T, Walker B, Phillips JK, Fejer R, Beck R. Hand-held dynamometry correlation with the gold standard isokinetic dynamometry: a systematic review. PM R. 2011 May;3(5):472-9. doi: 10.1016/j.pmrj.2010.10.025. PMID 21570036
- [Background] Andersen LB, Abrahamsen B, Dalgard C, Kyhl HB, Beck-Nielsen SS, Frost-Nielsen M, Jorgensen JS, Barington T, Christesen HT. Parity and tanned white skin as novel predictors of vitamin D status in early pregnancy: a population-based cohort study. Clin Endocrinol (Oxf). 2013 Sep;79(3):333-41. doi: 10.1111/cen.12147. Epub 2013 Jul 2. PMID 23305099
- [Background] Lykkedegn S, Beck-Nielsen SS, Sorensen GL, Andersen LB, Fruekilde PBN, Nielsen J, Kyhl HB, Joergensen JS, Husby S, Christesen HT. Vitamin D supplementation, cord 25-hydroxyvitamin D and birth weight: Findings from the Odense Child Cohort. Clin Nutr. 2017 Dec;36(6):1621-1627. doi: 10.1016/j.clnu.2016.10.008. Epub 2016 Oct 27. PMID 27817876
- [Background] Kyhl HB, Jensen TK, Barington T, Buhl S, Norberg LA, Jorgensen JS, Jensen DF, Christesen HT, Lamont RF, Husby S. The Odense Child Cohort: aims, design, and cohort profile. Paediatr Perinat Epidemiol. 2015 May;29(3):250-8. doi: 10.1111/ppe.12183. Epub 2015 Mar 10. PMID 25756293